CLINICAL TRIAL: NCT06956352
Title: Impact of Collaborative Care for Pregnant Women With Opioid Use Disorder in Low-Resource Obstetric Settings
Acronym: NEST
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Magee-Women's Research Institute (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Krans, MD, Associate Professor, University of Pittsburgh
Other Study IDs: STUDY24030140; R61DA061377 (NIH)
Record Dates: First submitted 2025-05-01; First posted 2025-05-04 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy; Postpartum Period; Opioid Use Disorder
Keywords: HEAL Inititative; HEAL; MOUD; OUD; Pregnancy; Postpartum; Substance
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adapted Collaborative Care Model (CCM): Person-centered, recovery supports.
  Interventions: Behavioral: Adapted Collaborative Care Model (CCM)
- Usual care: Usual, referral-based, care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Usual Care — Usual, referral-based, care.
  Groups: Usual care
Behavioral: Adapted Collaborative Care Model (CCM) — Person-centered, recovery supports.
  Groups: Adapted Collaborative Care Model (CCM)

SUMMARY:
The investigators seek to adapt a collaborative care model (CCM) for community-based, low-resource obstetric settings and to test the effects of this adapted CCM on health outcomes among Pregnant, postpartum, and parenting person (PPPP) with Opioid use disorder (OUD) and their families. To achieve this goal, investigators will conduct a nonrandomized, Type 1 hybrid implementation-effectiveness study across 3 community-based, low-resource obstetric sites in Northwest PA, a region with rates of maternal opioid-related diagnoses 4 times higher than national averages.

DETAILED DESCRIPTION:
Our central hypothesis is that person-centered, recovery supports, provided in the CCM will increase medication for OUD (MOUD) initiation and continuation, decrease overdose and reduce child removal rates among PPPP with OUD.

Specifically, investigators will:

1. Conduct an intervention adaptation project to adapt the Pregnancy and Women's Recovery Center (PWRC) CCM for rural and low-resource obstetric settings; and
2. Create a common data model to harmonize variables across data sources and data collection processes across study sites.

Investigators will also:

1. Evaluate the effects of the adapted PWRC CCM on outcomes among PPPP with OUD;
2. Determine if improvements in person-centered, recovery supports mediate the relationship between PWRC Community and outcomes using causal mediation methods; and
3. Identify PWRC Community adaptations that are associated with increased MOUD access, improved outcomes and that facilitate sustainability and scalability.

Research findings will:

1. provide high-quality evidence on how CCMs affect service delivery and health outcomes for PPPP with OUD,
2. inform stakeholders about ways to adapt CCMs for low-resource and rural healthcare settings, and
3. inform policymakers about the adaptations necessary to replicate these models widely.

ELIGIBILITY:
Inclusion Criteria:

(Stakeholder Participant)

1. 18 years or older
2. Providing care at participating obstetric site
3. English speaking

(Patient Participant)

1. 18 years or older
2. Receiving care at participating obstetric site
3. English speaking

Exclusion Criteria:

1. Unwillingness to have participation audio recorded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A core team of clinical providers at each obstetric site (i.e., nurse case manager, peer navigator, advanced practice provider, behavioral health provider, and lead obstetrician/gynecologist) have already committed to providing clinical care for the adapted CCM and participate in all stages of the research process. As such, they will not need to be recruited for participation.
  Maternal and child outcome data will be collected retrospectively from the EHR and individual patients will not be recruited to participate in the study. A small subset of pregnant women (n=50) who meet DSM-V criteria for OUD and who receive care at obstetric sites will be recruited for a one-time, semi-structured qualitative interview.
Sampling Method: Non-Probability Sample
Enrollment: 1350 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Patient Initiation of Medication for Opioid Use Disorder (MOUD) | During pregnancy (up to 40 weeks), up to 1 year post delivery
  Patient Initiation of Medication for Opioid Use Disorder (MOUD) as measured by total buprenorphine or methadone initiation in Electronic Health Record (EHR) and Medicaid claims data
Patient Duration of MOUD | During pregnancy (up to 40 weeks), up to 1 year post delivery
  Patient Duration of MOUD as measured by proportion of days' covered incorporating buprenorphine or methadone treatment in EHR and claims data
Patient Overdose | During pregnancy (up to 40 weeks), up to 1 year post delivery
  Patient Overdose as measured by total count of nonfatal or fatal overdose events in EHR and claims data
Patient child foster care placement | Delivery through 1 year postpartum
  Patient child foster care placement as measured by total child placements in foster care system according to child protective service data linked with Medicaid data
Patient utilization of well-child services | Delivery through 1 year postpartum
  Patient utilization of well-child services as measured by total well-child visits in EHR and claims data

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Krans, MD, Principal Investigator — University of Pittsburgh; Marian Jarlenski, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
HEAL Data Platform (HDP01418); NAHDAP data repository.
Time Frame: Before publishing and/or at the end of the study period with results.
Access Criteria: Public Access and Data Sharing Plan: A Public Access and Data Sharing Plan describes the plan for releasing Publications and sharing the Underlying Primary Data for an NIH HEAL Initiative Research Project.
URL: https://heal.nih.gov/data/complying-heal-data-sharing-policy